CLINICAL TRIAL: NCT02767505
Title: Bypass Equipoise Sleeve Trial (BEST); A Randomised Controlled Multicenter Trial Comparing Gastric Bypass and Sleeve Gastrectomy
Brief Title: Bypass Equipoise Sleeve Trial (BEST)
Acronym: BEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Ersta Hospital, Sweden (Other); Region Örebro County (Other); Kalmar County Hospital (Other); Lindesbergs Hospital (Unknown); Danderyd Hospital (Other); Skaraborg Hospital (Other Government); Sodertalje Hospital (Other); Östra Hospital (Other); Mora Hospital (Unknown); Torsby Hospital (Unknown); Stockholm South General Hospital (Other); Gävle Hospital (Other); Uppsala University Hospital (Other); Lycksele Hospital (Unknown); Falu Hospital (Other); Vrinnevi Hospital, Norrköping (Unknown); Capio S:t Görans Hospital (Unknown); Ljungby Hospital (Unknown); Sykehuset i Vestfold HF (Other); Gjövik Hospital, Norway (Unknown); GB Obesitas Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 478-15, version 5 2020-03-23
Record Dates: First submitted 2015-11-04; First posted 2016-05-10 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleeve gastrectomy (Experimental): Laparoscopic sleeve gastrectomy
  Interventions: Other: Sleeve gastrectomy
- Gastric bypass (Active Comparator): Laparoscopic Roux-en-Y gastric bypass
  Interventions: Other: gastric bypass

INTERVENTIONS:
Other: gastric bypass — Type of surgery: gastric bypass
  Arms: Gastric bypass
Other: Sleeve gastrectomy — Typ of surgery: sleeve gastrectomy
  Arms: Sleeve gastrectomy

SUMMARY:
This is nationwide registry-based randomised clinical multicenter trial in which patients will be randomised to gastric bypass (RYGB) or sleeve gastrectomy (SG). The co-primary endpoint are weight control over 5 years and the amount of severe adverse events. Additionally the investigators have predefined a number of secondary endpoints, and the trial has a sufficient number of patients to allow comparisons across subgroups.

DETAILED DESCRIPTION:
Follow-up of the patients will use the routines respectively for regular follow-up on the Scandinavian Obesity Surgery Registry (SOReg) after 6v, 1 year, 2 years, and after 5 years.

In order to evaluate if SG has advantages compared to the previous standard, the investigators want to examine whether SG operations are equivalent (non-inferiority) for weight loss and weight stability five years after surgery in comparison to RYGB, and if SG is associated with fewer long-term complications (superiority). The primary outcome measure emanates from assessment of long term weight management and the frequency of serious complications.

The unforeseen global Covid-19 pandemic resulted in that almost all elective benign surgery in Scandinavia was cancelled from March 2020. Thus, the pandemic had severe consequences on the recruitment to the BEST trial during 2020-2021.

During autumn of 2021 the BEST steering committee decided to perform an additional analysis of the power for primary endpoints.

Additional information (Courcoulas et al, JAMA Surg 2020 March; Howard et al, JAMA Surg 2021 Dec) revealed that the risk of any of the predefined substantial adverse events after bariatric surgery is higher than previously anticipated in the revised power calculation, i.e. >25% instead of 13%. These figures were confirmed in an analysis of real-world data from the bariatric national quality register SOReg in Sweden which registered all patients undergoing sleeve or bypass in Sweden since 2007.

An independent statistician performed the analysis based on information above, but also on 2-year data in BEST. In conclusion, it was stated:

Two post hoc power analyses were conducted based on the data from February 2022:

1. Weight reduction. In the protocol the following is stated "This sample size will also have >95% power to evaluate non-inferiority of 5% weight loss difference over 5 years between the two groups, assuming 15 kg standard deviation in weight loss over follow-up with two-sided 2.5% significance level.". The post hoc power calculation is based on the two-year follow up data where an average weight loss for all patients (both groups, N=1031) of 29.3 kg was attained with a Sd=21.6. Given a loss to follow up of 20% from 2 year follow up to the 5-year follow up the sample size is assumed to be (1031*0.80)/2=413 patients per group. With a non-inferiority level of 5 kg weight loss the power is found to be 90% if n=393 per group, and 95% if n=486 per group (https://www.sealedenvelope.com/power/continuous-noninferior/).
2. Substantial adverse events. This post hoc power calculation is for a superiority test where the rate is assumed to be 25% for the gastric bypass at 5 years and sleeve would have a 35% lower level, i e 25%*0.65=16.25%. Given a sample of n=413 per group the post hoc power will then be 87.5%.

Taking information above into account and in the interest of not prolonging inclusion period unnecessarily the trial steering committee took a decision to stop inclusion in BEST during spring 2022 (final date 31st of March). At termination of inclusion the number of participants that had been included and operated in BEST were 1752. The trial Data Safety and Monitoring Committee reviewed and supported the decision before termination of recruitment to the BEST trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35-50 kg/m2
* Ability to understand and decide on the merits of the study participation
* Accepted for bariatric surgery
* Must understand the information, and be able to make a decisions about participation in the study

Exclusion Criteria:

* Previous bariatric surgery, anti reflux surgery or other gastric surgery
* Moderate to severe reflux disease, Barretts oesophagus or known hiatus hernia >4 cm
* Unstable mental illness or other known contraindication to bariatric surgery.
* Planned significant surgery at the same time
* Inflammatory bowel disease
* ongoing drug or substance abuse
* not appropriate to randomise the patient, according to surgeon

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1752 (Actual)
Dates: Start 2015-09; Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 5 years
  Non-inferiority for SG is defined as < 5% weight difference
Serious adverse events | 5 years
  Superiority for SG is having 35% less serious (substantial) adverse events compared to RYGB

SECONDARY OUTCOMES:
Adverse events | 1, 2, 5 and 10 years
  General description of patterns of all adverse events
Weight loss | Baseline, 1, 2, 5 and 10 years
  Between baseline and 1 and 2 years
Number of patients with arterial cardiovascular events | Baseline, 1, 2, 5 and 10 years
  Composite of myocardial infarction+ stroke+ other occlusive arterial condition
Number of patients with venous event | Baseline, 1, 2, 5 and 10 years
  Composite of Deep vein thrombosis+ Pulmonary emboli+ other venous event
Number of patients with diabetes requiring drug treatment | Baseline, 1, 2, 5 and 10 years
  Development of diabetes measured as numbers of patients having a diabetes diagnosis and oral medication and injection therapy
Number of patients with a psychiatric morbidity | Baseline, 1, 2, 5 and 10 years
  Number of patients with a psychiatric morbidity
Number of patients with hypertension treatment | Baseline, 1, 2, 5 and 10 years
  Number of patients with hypertension treatment (any type of Medical treatment)
Number of patients diagnosed with a malignancy | Baseline, 1, 2, 5 and 10 years
  Number of patients diagnosed with a malignancy
Number of patients with dyslipidemia treatment | Baseline, 1, 2, 5 and 10 years
  Number of patients with diagnosis of dyslipidemia and on oral lipid lowering treatment
Weight in men and women | Baseline, 1, 2, 5 and 10 years
  Analyses of the primary outcome weight in men and women
serious adverse events in men and women | Baseline, 1, 2, 5 and 10 years
  Analyses of the primary outcome serious adverse events in men and women
Weight in patients with BMI >43 vs <43 kg/m2. | Baseline, 1, 2, 5 and 10 years
  Analyses of the primary outcome weight in patients with BMI >43 vs <43 kg/m2.
Serious adverse events in patients with BMI >43 vs <43 kg/m2 | Baseline, 1, 2, 5 and 10 years
  Analyses of the primary outcome serious adverse events in patients with BMI >43 vs <43 kg/m2.
Weight in patients aged 18-25 y, 25-50 y, or >50 y | Baseline, 1, 2, 5 and 10 years
  Analyses of the primary outcome weight in patients aged 18-25 y, 25-50 y, or >50 y
Serious adverse events in patients aged 18-25 y, 25-50 y, or >50 y | Baseline, 1, 2, 5 and 10 years
  Analyses of the primary outcome serious adverse events in patients aged 18-25 y, 25-50 y, or >50 y
Mineral nutritional status | Baseline, 1, 2, 5 and 10 years
  Serum concentrations of iron depots, zinc, magnesium, selenium and copper
Vitamin nutritional status | Baseline, 1, 2, 5 and 10 years
  Serum concentrations of vitamins (Vitamin B12, Vitamin D, Vitamin A, thiamin)
Serum concentrations of albumin | Baseline, 1, 2, 5 and 10 years
  Serum concentrations of Albumin
Changes in quality of Life assessed with EQ-5D | Baseline, 1, 2, 5 and 10 years
  Assessed with EQ-5D
Changes in quality of Life assessed with Obesity Problems (OP) | Baseline, 1, 2, 5 and 10 years
  Assessed with Obesity Problems (OP)
Changes in quality of Life assessed with Short Form-36 | Baseline, 1, 2, 5 and 10 years
  Assessed with SF-36
Alcohol consumption | 1, 2, 5 and 10 years
  Assessed by AUDIT
Gastro-esophageal reflux disease | 1, 2, 5 and 10 years
  Gastro-esophageal reflux disease is defined as present/ not present in at least one of following modalities: Questionnaire DeMeester score, 24h pH manometry and/or gastroscopy
Fracture incidence | 2, 5 and 10 years
  From clinical data and national registry
Bone density and body composition | 10 years
  Dual energy X-ray Absorptiometry (DEXA) in at least a subgroup of 500+500
Mortality and cause of death | 5, 10, 20 and 30 years
  National Cause of Death registry
Health care consumption, In hospital registry | 5, 10, 20 and 30 years
  Data from In hospital registry (Days in hospital)
Health care consumption, | 5, 10, 20 and 30 years
  Data from Outpatient registry ( number of visits)
Health care consumption | 5, 10, 20 and 30 years
  National drug registry (type of drug)
Development of co-morbidities from national registry data | 5, 10, 20, 30 years
  National stroke registry, National Cardiac registry, National Diabetes Registry, Cancer registry
Formal cost effective analysis | 5, 10 and 20 years
  Cost per quality-adjusted life-year and life-year)
Dietary intake | 1 and 10 years
  Questionnaire regarding food intake (E14x)
Eating patterns | 1 and 10 years
  Three Factor Eating Questionnaire (TFEQ)
Gastro-intestinal side effects | 1 and 10 years
  Questionnaire: Gastro-intestinal Symptom Rating Score (GSRS)
Dumping symptoms | 1 and 10 years
  Questionnaire: Dumping Symptom Rating Score (DSRS)
Adverse events | 30 days postop, 1, 2, 5 and 10 years
  Clinical data combined with national registry data
Peri-operative outcome, Complications | Up to 30 days postop
  Complications; Surgical (minor/major) and medical
Peri-operative outcome, surgical time | Up to 30 days postop
  surgical time (min)
Peri-operative outcome, sick leave | Up to 30 days postop
  sick leave (days)
Peri-operative outcome, length of stay | Up to 30 days postop
  length of stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Olbers, MD, PhD, Principal Investigator — Linköping University, Dept of BKV
Locations (21):
- Sentralsykehuset Vestfold, Tønsberg, Norway
- Sweden (20):
  - Falu Hospital, Falun
  - Gävle Hospital, Gävle
  - Östra Hospital, Gothenburg
  - Kalmar County Hospital, Kalmar
  - Lindesbergs Hospital, Lindesberg
  - Linköping University, Linköping
  - Ljungby Hospital, Ljungby
  - Lycksele Hospital, Lycksele
  - Mora Hospital, Mora
  - Vrinnevi Hospital, Norrköping, Norrköping
  - Örebro University Hospital, Örebro
  - GB Obesitas, Skåne
  - Skaraborgs Hospital, Skövde
  - Södertälje Hospital, Södertälje
  - Ersta Hospital, Stockholm
  - Danderyds Hospital, Stockholm
  - Capio S:t Görans Hospital, Stockholm
  - Stockholm South General Hospital, Stockholm
  - Torsby Hospital, Torsby
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hedberg S, Thorell A, Osterberg J, Peltonen M, Andersson E, Naslund E, Hertel JK, Svanevik M, Stenberg E, Neovius M, Naslund I, Wiren M, Ottosson J, Olbers T; BEST Study Group. Comparison of Sleeve Gastrectomy vs Roux-en-Y Gastric Bypass: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2353141. doi: 10.1001/jamanetworkopen.2023.53141. PMID 38289603
- [Derived] Hedberg S, Olbers T, Peltonen M, Osterberg J, Wiren M, Ottosson J, Thorell A; BEST study group. BEST: Bypass equipoise sleeve trial; rationale and design of a randomized, registry-based, multicenter trial comparing Roux-en-Y gastric bypass with sleeve gastrectomy. Contemp Clin Trials. 2019 Sep;84:105809. doi: 10.1016/j.cct.2019.07.001. Epub 2019 Jul 4. PMID 31279778